CLINICAL TRIAL: NCT05575570
Title: Pre-emptive Abdominal Aortic Aneurysm Sac Embolization During Endovascular Abdominal Aortic Repair for Infrarenal Abdominal Aortic Aneurysm - Randomized Study
Brief Title: Pre-emptive Abdominal Aortic Aneurysm Sac Embolization During EVAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Stevo Duvnjak, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-22000209
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture
Keywords: AAA; Embolization; Endoleak; sac regression
MeSH Terms: conditions — Endoleak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-emptive AAA sac embolization (Active Comparator)
  Interventions: Device: EVAR
- No pre-emtive AAA sac embolization (Sham Comparator)
  Interventions: Device: EVAR

INTERVENTIONS:
Device: EVAR — EVAR stent graft and embolization material CE marked.

SUMMARY:
Pre-emptive abdominal aortic aneurysm sac embolization during endovascular abdominal aortic repair for infrarenal abdominal aortic aneurysm - Randomized study

DETAILED DESCRIPTION:
In all 124 patients will be included, 62 in each group.

The first group (62 patients) with pre-emptive AAA sac embolization during EVAR and the control group consisted of 62 patients without pre-emptive AAA sac embolization.

The primary goal is to investigate AAA shrinkage/diameter changes in the pre-emptive embolization group compared with the non-embolization group. Further, to investigate all endoleaks and secondary interventions during the follow-up and any difference between groups and correlation if any with pre-emptive embolization.

Demographic, comorbidities, antiplatelet and anticoagulation drugs, AAA characteristics, patent lumbal and inferior mesenteric artery, intervention characteristics and follow-up data will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with 55mm (male) or 50 mm (female) AAA, available for EVAR
* > 18 year old

Exclusion Criteria:

* Not accept to participate
* Ruptured AAA
* Outside for instruction for the use EVAR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
AAA diameter and volume changes/sac regression during follow-up, measurement on control CT and/or ultrasound after EVAR. | 5 years
  Sac regression uses the centerline reconstruction to compare the baseline CT aorta scanning and AAA diameter measurement - maximal AAA diameter in millimetres (mm).
  Further, total volume measurement in (ml) of AAA and sac changes during the follow-up comparing the index CT scan with control CT or ultrasound scanning.
AAA diameter and volume changes/sac regression during follow-up, measurement on control CT with automatic volume software program | 3 years
  1. Automatic software measured the maximal AAA diameter in millimetres (mm) on index CT and follow-up control scanning. The same technique and measurement points will be used. Specialised software dedicated to AAA maximal diameter will be used.
  2. Automatic software measurement of total volume of AAA in millilitres (ml) on index CT scanning and on control CT scanning. Specialised software will perform measurement and volumetry expressed in millilitres (ml).

SECONDARY OUTCOMES:
Secondary interventions, endovascular secondary interventions( additional embolization, a new stent graft deployment etc) | 5 years
  The type of secondary interventions, incidence, time to secondary intervention, and the outcome will be recorded and analysed.
Endoleak type 2 incidence, on control CT and ultrasound scanning | 5 years
  Incidence of endoleak type 2 and other endoleak will be noted and analysed.

IPD SHARING:
Plan to Share IPD: No